CLINICAL TRIAL: NCT00803530
Title: Phase II Multicenter Study of Association of Arsenic Trioxide (ATO) and Ascorbic Acid in Myelodysplastic Syndromes
Brief Title: Study of Association of Arsenic Trioxide (ATO) and Ascorbic Acid in Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: difficulties of enrollement
Sponsor: Fondazione Italiana Sindromi Mielodisplastiche-ETS (Other)
Collaborators: Centro di Riferimento per l'Epidemiologia e la Prev. Oncologica Piemonte (Other)
Responsible Party: Alessandro Levis, Azienda Ospedaliera SS Antonio e Biagio, Alessandria.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AISSM02A; EudracT Number 2005-001321-28
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Myelodysplastic Syndromes
Keywords: myelodysplastic syndromes; arsenic trioxide; ascorbic acid
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Loading phase (week 1): ATO 0.3 mg/Kg/die for 5 consecutive days.
  * Subsequent phase (from week 2 to week 16): ATO 0.25 mg/kg twice a week (day 2 and 5 of every week).
  * Ascorbic acid 1000 mg IV within 30 minutes after each arsenic trioxide infusion for 16 consecutive weeks.
  Interventions: Drug: ATO + Ascorbic acid

INTERVENTIONS:
Drug: ATO + Ascorbic acid — ATO will be diluted in 250 ml of normal saline solution at a dosage of 0.3 mg/Kg during the first week of therapy and at a dosage of 0.25 mg/Kg during the subsequent weeks (week 2 to 16), and administered intravenously over a 1-2 hour period.
  The dose of ascorbic acid will be 1000 mg in 100 cc D5W or normal saline solution (NaCl 0.9 %) (protected from light and air) administered as an IV infusion over 15 to 30 minutes. The dosing solution is not to be mixed with any alkaline solution.

SUMMARY:
This is a prospective, multicenter phase II trial designed to evaluate the safety and activity of the combination of association of arsenic trioxide (ATO) and ascorbic acid in patients with myelodysplastic syndromes

ELIGIBILITY:
Inclusion Criteria:

1. Patients affected by myelodysplastic syndromes, entering in one of the following groups:

   1. Myelodysplastic syndromes independent of WHO diagnostic classification (43) and IPSS prognostic score (2), when present at least one of the following abnormalities:

      * 3q26 chromosome rearrangement.
      * High EVI-1 transcript levels.
   2. Myelodysplastic syndromes without excess of blasts (non-RAEB patients) at low or intermediate-1 score risk according to the IPSS (2), as a second line treatment option, after a failure to the first line treatment with erythropoietin +/- G-CSF, immunosuppressive therapy, or other initial treatment modality.
   3. Non RAEB patients at intermediate-2 or high risk score or RAEB patients at any prognostic score, who are non candidate to treatment with conventional chemotherapy regimens.
2. Presence of one ore more cytopenias characterised by one ore more of the following elements:

   * Transfusions dependence.
   * Hb< 11 gr/dl
   * Platelet count < 50x109/L
   * Absolute neutrophil count < .5x109/L.
3. ECOG Performance status ≤ 2.
4. Aged from 18 to 80.
5. Life expectancy > 4 months.
6. Creatinine level < 1.5 mg/dl.
7. Liver function tests, including ASL-ALT-alkaline phosphatase lower than 3xULN
8. No previous treatment with chemotherapy, growth factors, cytokines or other experimental treatment within 4 weeks of starting treatment.
9. No history of clinically significant cardiac disease, including congestive heart failure.
10. Cytogenetic evaluation available.
11. Sending of both peripheral blood and bone marrow sample to the central laboratory for EVI-1 rearrangement evaluation.
12. Written Informed consent.

Exclusion Criteria:

1. Patients affected by myelodysplastic syndromes entering in categories other than those foreseen by inclusion criteria point 1.
2. Absence of cytopenia defined as the contemporarily presence of all the following conditions: a) no transfusion need; b) Hb > 11 gr/dl; c) platelet count > 50x109/L; d) absolute neutrophil count > .5x109/L.
3. All patients that might be candidate to allogenic stem cell transplantation.
4. Patients that might be candidate to a first line immunosuppressive therapy.
5. ECOG Performance status > 2.
6. Age lower than 18 or higher then 80.
7. Life expectancy < 4 months.
8. Creatinine level > 1.5 mg/dl.
9. Liver function tests, including ASL-ALT-alkaline phosphatase higher than 3xULN
10. Treatment with chemotherapy, growth factors, cytokines or other experimental treatment within 4 weeks of starting treatment.
11. Clinically significant cardiac disease, including congestive heart failure, rhythm abnormalities, QT time > 460m/s, or need of anti-arrhythmic drugs.
12. Concurrent co-morbid medical condition which might exclude administration of therapy, as judged by individual investigator.
13. Absence of cytogenetic evaluation.
14. Participation at same time in another study in which investigational drugs are used.
15. Absence of written Informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
TO evaluate the erythroid response rate (major), according to the International Working Group (IWG) criteria (42) after four months of treatment with the association of ATO and ascorbic acid. | 16 mounths

SECONDARY OUTCOMES:
To evaluate platelets and granulocyte response according to the International Working Group (IWG) criteria (42) after four months of treatment with the association of ATO and ascorbic acid | 16 mounths

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Levis, MD, Study Director — S.O.C. di Ematologia, Azienda Ospedaliera SS Antonio e Biagio, Alessandria. Via Venezia 18 - 15100 - Alessandria
Locations (13):
- Italy (13):
  - Ospedale SS Antonio, Biagio e Cesare Arrigo, Alessandria
  - Ospedale Cardinal Massaia, Asti
  - Spedali Civili, Brescia
  - Ospedale Maggiore, Chieri
  - Ospedale civico di Chivasso, Chivasso (TO)
  - Ospedale Santa Croce e Carle, Cuneo
  - AOS San Gerardo de' Tintori, Monza
  - Università Avogadro Divisione di Ematologia, Novara
  - Ospedale San Luigi Gonzaga Divisione di Ematologia, Orbassano (TO)
  - Azienda Ospedaliera Perugia, Perugia
  - Ospedale San Giovanbni Battista-Molinette, Torino
  - Ospedale San Giovanni Battista -Molinette, Torino
  - Ospedale San Bortolo, Vicenza

REFERENCES:
- [Derived] Galimberti S, Guerrini F, Salvi F, Petrini I, Gioia D, Messa E, Palumbo GA, Cilloni D, Petrini M, Levis A. Arsenic trioxide and ascorbic acid interfere with the BCL2 family genes in patients with myelodysplastic syndromes: an ex-vivo study. J Hematol Oncol. 2012 Sep 10;5:53. doi: 10.1186/1756-8722-5-53. PMID 22964015